CLINICAL TRIAL: NCT03615872
Title: Evaluation of Patient Satisfaction With Pessary in the Treatment of Genital Prolapse
Brief Title: Pessary Satisfaction Criteria for Urogenital Prolapse
Acronym: PeSaCUP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A00004-51
Record Dates: First submitted 2018-07-16; First posted 2018-08-06 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-08

CONDITIONS: Genital Prolapse; Pessary; Satisfaction
Keywords: quality of life; efficiency
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: pessary use — evaluation of satisfaction of pessary use in case of symptomatic genital prolapse

SUMMARY:
Genital prolapse is a common pathology with a prevalence ranging from 2.9 to 11.4% or 31.8% to 97.7%, depending on whether a questionnaire or clinical examination is used. The use of pessary in the treatment of prolapse remains discussed despite a satisfaction rate of 50 to 80% in the literature and a minimal complications rate.

The main objective of this study is to assess the satisfaction of patients carrying a pessary in the first year after the laying.

DETAILED DESCRIPTION:
This is a prospective observational cohort conducted at the Universitary hospital of Caen over a total period of 5 years.

Patients with a symptomatic genital prolapse will all be offered the installation of a pessary. If they agree to participate in the study, they will be asked to respond to validated questionnaires: symptom questionnaires (PFDI-20, ICIQ-SF, USP), a sexuality questionnaire (PISQ-12), a quality of life questionnaire (PFIQ-7, BIS) and Satisfaction (PGI-I), several times: Before the installation of the pessary, at one month, at 6 months, then annually over 5 years

ELIGIBILITY:
Inclusion Criteria:

* The research protocol will be proposed to all patients with a symptomatic genital prolapse, over 18 years of age, who speak French and who agree to participate in this study
* Prolapse defined according to the International Classification POP-Q-.

Exclusion Criteria:

* Minors under 18 years of age
* Pregnant or lactating women
* Women Not speaking French (the good understanding of French is necessary to answer questionnaires and for informed information)
* Women unable to understand due to cognitive impairment or degenerative disease (dementia/ Alzheimer's disease)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research protocol will be proposed to all patients with a symptomatic genital prolapse
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Patient SATISFACTION assessed by the PGI-I score (Patient Global Impression of Improvement) in the first year after the installation of a pessary | 1 year
  The PGI-I score was developed and validated to quantify the effect of urinary incontinence or prolapse treatments

SECONDARY OUTCOMES:
Patient SATISFACTION assessed by the PGI-I score (Patient Global Impression of Improvement) every year for five years after the installation of a pessary | 1 to 5 years
  The PGI-I score was developed and validated to quantify the effect of urinary incontinence or prolapse treatments
EFFICACY of pessary on genital symptoms assessed by the Pelvic Floor Distress Inventory (PFDI-20) questionnaire before and after the installation of the pessary. | at 1 year, then every year for 5 years
  This score was developped to evaluate the genital, anorectal and urinary symptoms related to genital prolapse
EFFICACY of pessary on urinary symptoms assessed by the International Consultation of Incontinence Questionnaire-Short Form (ICIQ-UI SF) and the Urinary Symptom Profile score (USP) before and after the installation of the pessary. | at 1 year, then every year for 5 years
  These scores are self-questionnaires specifically validated to evaluate urinary incontinence and urinary tract dysfunctions
Sexual impact of pessary assessed by the Pelvic organ prolapse urinary Incontinence Sexual Questionnaire (PISQ-12) | at 1 year, then every year for 5 years
  Evaluation of the PISQ-12 score after the installation of a pessary. This score was developped specifically to evaluate sexual troubles in case of genital prolapse
QUALITY OF LIFE assessed by the Pelvic Floor Impact Questionnaire (PFIQ-7) before and after the installation of the pessary | at 1 year, then every year for 5 years
  The PFIQ-7 was developped to evaluate the impact of the symptoms on the quality of life
INVESTIGATE the impact of age on the removal or expulsion of pessary | 1 year to 5 years
  Impact of age (years) on treatment failure (removal or expulsion of pessary)
INVESTIGATE the impact of menopausal status on the removal or expulsion of pessary | 1 year to 5 years
  Impact of menopausal status (yes/no) on treatment failure (removal or expulsion of pessary)
INVESTIGATE the impact of weight on the removal or expulsion of pessary | 1 year to 5 years
  Impact of weight (Kg) on treatment failure (removal or expulsion of pessary)
INVESTIGATE the impact of hysterectomy history on the removal or expulsion of pessary | 1 year to 5 years
  Impact of hysterectomy history (yes/no) on the removal or expulsion of pessary
INVESTIGATE the impact of prolapse surgery history on the removal or expulsion of pessary | 1 year to 5 years
  Impact of prolapse surgery history (yes/no) on the removal or expulsion of pessary
INVESTIGATE the impact of the prolapse stage of on the removal or expulsion of pessary | 1 year to 5 years
  Impact of the prolapse stage (assessed by the validated POP-Q classification) of on the removal or expulsion of pessary. The stage of prolapse is ranged from 1 to 4 in the POP-Q classification
Complications of pessary use reported by their rate | 1 to 5 years
  Rate of complications related to the use of a pessary (frequencies)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Cecile PIZZOFERRATO, MD, Principal Investigator — Universitary Hospital of Caen
Locations (1):
- Pizzoferato, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided
The IPD will be shared with the researchers working with me for the study, i.e. Dr Villot and Miss Renouf

REFERENCES:
- [Background] Cundiff GW, Amundsen CL, Bent AE, Coates KW, Schaffer JI, Strohbehn K, Handa VL. The PESSRI study: symptom relief outcomes of a randomized crossover trial of the ring and Gellhorn pessaries. Am J Obstet Gynecol. 2007 Apr;196(4):405.e1-8. doi: 10.1016/j.ajog.2007.02.018. PMID 17403437
- [Background] Clemons JL, Aguilar VC, Tillinghast TA, Jackson ND, Myers DL. Patient satisfaction and changes in prolapse and urinary symptoms in women who were fitted successfully with a pessary for pelvic organ prolapse. Am J Obstet Gynecol. 2004 Apr;190(4):1025-9. doi: 10.1016/j.ajog.2003.10.711. PMID 15118635
- [Background] Patel M, Mellen C, O'Sullivan DM, LaSala CA. Impact of pessary use on prolapse symptoms, quality of life, and body image. Am J Obstet Gynecol. 2010 May;202(5):499.e1-4. doi: 10.1016/j.ajog.2010.01.019. Epub 2010 Feb 20. PMID 20171608
- [Background] Lone F, Thakar R, Sultan AH, Karamalis G. A 5-year prospective study of vaginal pessary use for pelvic organ prolapse. Int J Gynaecol Obstet. 2011 Jul;114(1):56-9. doi: 10.1016/j.ijgo.2011.02.006. Epub 2011 May 14. PMID 21575953
- [Background] Clemons JL, Aguilar VC, Sokol ER, Jackson ND, Myers DL. Patient characteristics that are associated with continued pessary use versus surgery after 1 year. Am J Obstet Gynecol. 2004 Jul;191(1):159-64. doi: 10.1016/j.ajog.2004.04.048. PMID 15295358
- [Background] Panman CM, Wiegersma M, Kollen BJ, Burger H, Berger MY, Dekker JH. Predictors of unsuccessful pessary fitting in women with prolapse: a cross-sectional study in general practice. Int Urogynecol J. 2017 Feb;28(2):307-313. doi: 10.1007/s00192-016-3107-4. Epub 2016 Aug 15. PMID 27525693
- [Background] Markle D, Skoczylas L, Goldsmith C, Noblett K. Patient characteristics associated with a successful pessary fitting. Female Pelvic Med Reconstr Surg. 2011 Sep;17(5):249-52. doi: 10.1097/SPV.0b013e31822f00ae. PMID 22453110
- [Background] Mutone MF, Terry C, Hale DS, Benson JT. Factors which influence the short-term success of pessary management of pelvic organ prolapse. Am J Obstet Gynecol. 2005 Jul;193(1):89-94. doi: 10.1016/j.ajog.2004.12.012. PMID 16021064
- [Background] Geoffrion R, Zhang T, Lee T, Cundiff GW. Clinical characteristics associated with unsuccessful pessary fitting outcomes. Female Pelvic Med Reconstr Surg. 2013 Nov-Dec;19(6):339-45. doi: 10.1097/SPV.0b013e3182a26174. PMID 24165447
- [Background] Kuhn A, Bapst D, Stadlmayr W, Vits K, Mueller MD. Sexual and organ function in patients with symptomatic prolapse: are pessaries helpful? Fertil Steril. 2009 May;91(5):1914-8. doi: 10.1016/j.fertnstert.2008.02.142. Epub 2008 Apr 14. PMID 18410935
- [Background] Jelovsek JE, Barber MD. Women seeking treatment for advanced pelvic organ prolapse have decreased body image and quality of life. Am J Obstet Gynecol. 2006 May;194(5):1455-61. doi: 10.1016/j.ajog.2006.01.060. PMID 16647928